CLINICAL TRIAL: NCT07078981
Title: Assessing Determinants of Headway in Evaluating Risk of Adhesion: the ADHERE Study
Brief Title: Adhesion Prevention in ASBO Surgery Using 4DryField® PH
Acronym: ADHERE
Status: Not yet recruiting | Type: Observational
Sponsor: Alessio Giordano (Other)
Collaborators: PlantTec Medical GmbH (Unknown)
Responsible Party: Sponsor-Investigator, Alessio Giordano, MD, General Surgeon, Azienda Sanitaria di Firenze
Organization: Azienda Sanitaria di Firenze (Other)
Other Study IDs: ADHERE2025
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Adhesive Small Bowel Obstruction; Postoperative Abdominal Adhesions; Bowel Obstruction; Abdominal Surgery Complications
Keywords: adhesion; obstruction; acute abdomen; emergency surgery; 4DryField; adhesiolysis; antiadhesion barrier; ASBO; abdominal surgery; peritoneal adhesion
MeSH Terms: conditions — Intestinal Obstruction; Tissue Adhesions; Bites and Stings; Abdomen, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antiadhesion Group: Patients undergoing surgery for ASBO who receive intraoperative 4DryField® PH application.
- No Antiadhesion Group: Patients undergoing surgery for ASBO without use of any antiadhesion agent.

SUMMARY:
Post-surgical adhesions occur in up to 90% of abdominal surgeries, often leading to complications like adhesive small bowel obstruction (ASBO) and chronic pain. They result from imbalanced healing processes influenced by growth factors, fibroblast activity, and genetic predispositions. While surgery can relieve ASBO, it frequently causes new adhesions, with recurrence rates up to 40%. Anti-adhesion barriers, such as the starch-based 4DryField® PH, form a temporary gel barrier to support healing. Though promising, its role in preventing ASBO recurrence is not well studied. This study evaluates whether intra-operative use of 4DryField® PH reduces ASBO recurrence over 12 months and compares perioperative outcomes in treated vs. untreated patients.

DETAILED DESCRIPTION:
Post-surgical adhesions are a common complication of abdominal surgery, with an occurrence rate of approximately 79-90%, leading to significant morbidity such as adhesive small bowel obstruction (ASBO) and chronic pain (1,2). These adhesions result from increased extracellular matrix production, reduced fibrinolytic activity, and the influence of growth factors like TGF-beta and VEGF, along with fibroblast proliferation(1). Genetic predispositions-affecting pathways such as TGF-β, VEGF, PAI-1, MMPs, and various pro-inflammatory cytokines-may increase the risk of adhesion formation(2-5).

Surgical management of ASBO resolves acute symptoms but often exacerbates the underlying issue by inducing further peritoneal trauma. Recurrence rates remain high-reported in up to 40% of patients-and complications from repeated adhesiolysis include increased operative time, bowel injury, and postoperative morbidity(6).

Various strategies have been explored in different surgical fields to prevent adhesion formation, including the use of physical antiadhesion barriers(7-9). Among these, 4DryField® PH, a plant-derived starch powder, has been shown to be safe and effective in clinical and experimental studies(8,10). When hydrated with saline, the powder forms a biocompatible gel that acts as a temporary barrier to physically separate traumatized serosal surfaces and allow for proper mesothelial regeneration.

Although the use of 4DryField® PH has been studied in different settings, there is limited prospective evidence evaluating its role in preventing recurrence of ASBO.

The present study aims to fill this gap by assessing whether intraoperative application of 4DryField® PH during surgery for ASBO reduces the recurrence rate during a 12-month follow-up, and by comparing perioperative outcomes between treated and untreated patients.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

* Undergoing surgical treatment for adhesive small bowel obstruction (ASBO)
* Ability and willingness to provide informed consent
* Willingness to adhere to follow-up visits

Exclusion Criteria:

* Presence of peritonitis
* Intra-abdominal active malignancy
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing surgery for adhesive small bowel obstruction (ASBO), including those with or without application of an antiadhesion agent, in real-world clinical settings.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of adhesive small bowel obstruction (ASBO) within 12 months | 12 months post-surgery
  Percentage of patients who experience a recurrence of adhesive small bowel obstruction (ASBO), based on clinical symptoms and imaging findings, during the 12-month follow-up period. Recurrence is defined by standardized clinical criteria (e.g. intermittent pain, nausea, vomiting, bowel obstruction symptoms) with or without radiological confirmation.

SECONDARY OUTCOMES:
Postoperative complications within 90 days | 90 days post-surgery
  Incidence and type of postoperative complications occurring within 90 days after surgery, classified according to Clavien-Dindo classification.

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared. Data collected in this study will be used solely for the purposes described in the protocol and will not be made available to other researchers.

REFERENCES:
- [Result] Ahmad M, Crescenti F. Significant Adhesion Reduction with 4DryField PH after Release of Adhesive Small Bowel Obstruction. Surg J (N Y). 2019 May 10;5(1):e28-e34. doi: 10.1055/s-0039-1687857. eCollection 2019 Jan. PMID 31093531
- [Result] Lorentzen L, Oines MN, Oma E, Jensen KK, Jorgensen LN. Recurrence After Operative Treatment of Adhesive Small-Bowel Obstruction. J Gastrointest Surg. 2018 Feb;22(2):329-334. doi: 10.1007/s11605-017-3604-x. Epub 2017 Oct 13. PMID 29030779
- [Result] Awonuga AO, Fletcher NM, Saed GM, Diamond MP. Postoperative adhesion development following cesarean and open intra-abdominal gynecological operations: a review. Reprod Sci. 2011 Dec;18(12):1166-85. doi: 10.1177/1933719111414206. Epub 2011 Jul 20. PMID 21775773
- See also: Related Info — https://www.aou-careggi.toscana.it/